CLINICAL TRIAL: NCT02356081
Title: eSMART: Randomised Controlled Trial to Evaluate Electronic Symptom Management Using the Advanced Symptom Management System (ASyMS) Remote Technology for Patients With Cancers
Brief Title: eSMART Trial to Evaluate ASyMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louise McKean (Other)
Collaborators: University College Dublin (Other); King's College London (Other); University of California, San Francisco (Other); University of Athens (Other); Medical University of Vienna (Other); University of Dundee (Other); European Cancer Patient Coalition (ECPC) (Unknown); Docobo Ltd. (Industry); University of Surrey (Other); Sykehuset Innlandet HF (Other)
Responsible Party: Sponsor-Investigator, Louise McKean, Solicitor, University of Strathclyde
Organization: University of Strathclyde (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CRC331
Record Dates: First submitted 2015-01-26; First posted 2015-02-05 (Estimated); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ASyMS intervention Group (Experimental): Patients in the intervention group will be instructed to use the ASyMS intervention once daily (and whenever they feel unwell) for up to 6 cycles of chemotherapy treatment.
  Interventions: Other: ASyMS intervention Group
- Control Group (No Intervention): Patients in the control group will receive standard care as is currently available at their clinical site.

INTERVENTIONS:
Other: ASyMS intervention Group — ASyMS is a mobile phone-based remote-monitoring system that enables the 'real-time' monitoring of patients' symptoms through use of a patient-reported outcome measure (PROM)
  Arms: ASyMS intervention Group

SUMMARY:
Chemotherapy may cause distressing symptoms which can impact on patients' quality of life. Chemotherapy is frequently given on an outpatient basis therefore patients are often required to manage the symptoms they experience at home without direct supervision from healthcare professionals. This study aims to evaluate the impact of a mobile phone based, remote monitoring, symptom management system (ASyMS) on the delivery of care to people with nonmetastatic breast, colorectal or haematological cancer during chemotherapy and for one year following treatment. The study aims to compare a number of outcomes of patients using the ASyMS intervention with outcomes of patients who receive normal care at their hospital. For up to 6 cycles of chemotherapy treatment, once a day and any other time they feel unwell, patients allocated to the mobile phone group will enter information on the phone regarding any symptoms they are experiencing, take their temperature and enter this on the phone. The information is sent via secure connection to a computer, which assesses the information and sends an alert to their health care professional in the hospital, who will call the patient at home if the patient has reported problematic symptoms. Patients in the normal care group will receive care as normal at their hospital. Both groups of patients will be asked to complete a series of questionnaires before they start treatment, after each chemotherapy cycle (for a maximum of 6 cycles) and at 3 monthly intervals for up to one year thereafter (a subset of patients will also be asked to complete midcycle symptom assessments). The study will also evaluate the cost benefit of ASyMS, assess changes in clinical practice as a result of ASyMS and develop a predictive risk model (statistical model) for use in future care of patients receiving chemotherapy for these cancers. This multicentre study is taking place across a number of European countries.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with breast cancer, colorectal cancer, or haematological malignancies (i.e. HD or NHL).
* Scheduled to receive first-line cytotoxic chemotherapy.
* Scheduled to receive 2-, 3- or 4-weekly chemotherapy protocols (i.e. chemotherapy administered at repeated cycles of 14, 21 or 28 days, respectively).
* Planned to receive a minimum of 3 chemotherapy cycles.
* Deemed physically/psychologically fit to participate in the study by a member of the multidisciplinary team.
* Able to understand and communicate in the respective language.

Exclusion Criteria:

* Patients with breast cancer or colorectal cancer with a distant metastasis, i.e. stage IV disease as defined by the TNM/UICC, (at the start of their chemotherapy treatment).
* Patients with a haematological malignancy (HD or NHL), who have B symptoms, (at the start of their chemotherapy treatment).
* Scheduled to receive concurrent radiotherapy during chemotherapy treatment.
* Scheduled to receive weekly chemotherapy protocols. Also, patients who shift from a 2-, 3- or 4-weekly protocol to a weekly protocol during chemotherapy will be excluded from further participation in the study.
* Diagnosed with the same type of cancer (i.e. where relapse has occurred) AND/OR another type of cancer (the only exception non-melanoma skin cancer) within the 5 years prior to recruitment to the study.
* Received chemotherapy treatment for any medical reason within the last 5 years, unless this is chemoradiation for colorectal cancer.
* Unable to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 829 (Actual)
Dates: Start 2015-02; Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Memorial Symptom Assessment Scale (MSAS) | At the end of each cycle of chemotherapy (each cycle can be either 14, 21 or 28 days long) for up to a maximum of 6 cycles of chemotherapy.
  The MSAS is a multidimensional selfreport questionnaire that evaluates 32 physical and psychological symptoms according to their frequency, severity and distress/bother to the person in the past week.

SECONDARY OUTCOMES:
Memorial Symptom Assessment Scale (MSAS) | At the halfway point during each cycle of chemotherapy (each cycle can be wither 14, 21 or 28 days long) for up to a maximum of 6 cycles of chemotherapy and/or at 3 monthly intervals for up to one year following a maximum of 6 cycles of chemotherapy.
  The MSAS is a multidimensional self-report questionnaire that evaluates 32 physical and psychological symptoms according to their frequency, severity and distress/bother to the person in the past week.
Functional Assessment of Cancer Therapy General (FACT-G) | At the end of each cycle of chemotherapy (each cycle can be either 14, 21 or 28 days long) for up to a maximum of 6 cycles of chemotherapy and/or at 3 monthly intervals for up to one year following a maximum of 6 cycles of chemotherapy.
  during active chemotherapy and/or at the 1 year follow-up
Supportive Care Needs Survey Short Form | At the end of each cycle of chemotherapy (each cycle can be either 14, 21 or 28 days long) for up to a maximum of 6 cycles of chemotherapy and/or at 3 monthly intervals for up to one year following a maximum of 6 cycles of chemotherapy.
  The 34-item instrument measures supportive care needs in five domains: health system and information, psychological needs, physical and daily living, patient care and support, and sexual-related.
State-Trait Anxiety Inventory-Revised | At the end of each cycle of chemotherapy (each cycle can be either 14, 21 or 28 days long) for up to a maximum of 6 cycles of chemotherapy and/or at 3 monthly intervals for up to one year following a maximum of 6 cycles of chemotherapy.
  The STAI-R is a 40-item measure of two types of anxiety - state anxiety (anxiety about an event), and trait anxiety (anxiety level as a personal characteristic). The State Anxiety scale assesses intensity of current feelings "at this moment". The Trait Anxiety scale assesses frequency of feelings 'in general'.
Communication and Attitudinal Self-Efficacy scale for cancer | At the end of each cycle of chemotherapy (each cycle can be either 14, 21 or 28 days long) for up to a maximum of 6 cycles of chemotherapy and/or at 3 monthly intervals for up to one year following a maximum of 6 cycles of chemotherapy.
  A 12-item measure of cancer patients' confidence and ability to engage in their self-care (i.e. self-efficacy) contributing to 3 dimensions (maintaining a positive attitude, understanding and participating in care, seeking and obtaining information).
Work Limitations Questionnaire | At the end of each cycle of chemotherapy (each cycle can be either 14, 21 or 28 days long) for up to a maximum of 6 cycles of chemotherapy and/or at 3 monthly intervals for up to one year following a maximum of 6 cycles of chemotherapy.
  A 25-item measure corresponding to 4 dimensions: time management; physical; mental/interpersonal; output demands). This was only completed by those individuals who were working.

OTHER OUTCOMES:
EuroQol 5-Dimensions combined with the Client Services Receipt Inventory | At the end of each cycle of chemotherapy (each cycle can be either 14, 21 or 28 days long) for up to a maximum of 6 cycles of chemotherapy and/or at 3 monthly intervals for up to one year following a maximum of 6 cycles of chemotherapy.
  To evaluate the cost-effectiveness of the intervention for the management of chemotherapy-related symptoms
Changes in clinical practice as a result of the intervention | Baseline and immediately after the intervention
  Exploring experiences of an anticipatory and preventative model of care
Predictive Risk Models (PRMs) to predict patients' chemotherapy-related symptoms by combining demographic, clinical, social and health service data collected from previous studies, as well as the current study, to inform the predictions made. | Daily throughout each cycle of chemotherapy (each cycle can be either 14, 21 or 28 days long) for up to a maximum of 6 cycles of chemotherapy.
  To move beyond traditional approaches to manage symptoms in oncology patients receiving chemotherapy to more tailored and anticipatory approaches.

CONTACTS AND LOCATIONS:
Overall Officials: Roma Maguire, Principal Investigator — University of Strathclyde
Locations (11):
- Medical University Vienna Comprehensive Cancer Center, Vienna, Austria
- Greece (3):
  - Agioi Anargiri Cancer Hospital, Athens
  - Air Force General Hospital, Athens
  - Metropolitan Hospital, Athens
- Ireland (2):
  - St James's Hospital, Dublin
  - St Vincent's Healthcare Group, Dublin
- Innlandet Hospital Trust, Lillehammer, Norway
- United Kingdom (4):
  - Guy's and St Thomas' NHS Foundation Trust, London
  - St George's Healthcare Trust, London
  - University College London, London
  - Mount Vernon Cancer Centre, Northwood

REFERENCES:
- [Derived] McCann L, Lewis L, Oduntan O, Harris J, Darley A, Berg GV, Lubowitzki S, Cheevers K, Miller M, Armes J, Ream E, Fox P, Furlong EP, Gaiger A, Kotronoulas G, Patiraki E, Katsaragakis S, McCrone P, Miaskowski C, Cardone A, Orr D, Flowerday A, Skene S, Moore M, De Souza N, Donnan P, Maguire R. Patients' and Clinicians' Experiences Using a Real-Time Remote Monitoring System for Chemotherapy Symptom Management (ASyMS): Qualitative Study. J Med Internet Res. 2024 Dec 3;26:e53834. doi: 10.2196/53834. PMID 39626227
- [Derived] Miller M, McCann L, Lewis L, Miaskowski C, Ream E, Darley A, Harris J, Kotronoulas G, V Berg G, Lubowitzki S, Armes J, Patiraki E, Furlong E, Fox P, Gaiger A, Cardone A, Orr D, Flowerday A, Katsaragakis S, Skene S, Moore M, McCrone P, De Souza N, Donnan PT, Maguire R. Patients' and Clinicians' Perceptions of the Clinical Utility of Predictive Risk Models for Chemotherapy-Related Symptom Management: Qualitative Exploration Using Focus Groups and Interviews. J Med Internet Res. 2024 Jun 20;26:e49309. doi: 10.2196/49309. PMID 38901021
- [Derived] Maguire R, McCann L, Kotronoulas G, Kearney N, Ream E, Armes J, Patiraki E, Furlong E, Fox P, Gaiger A, McCrone P, Berg G, Miaskowski C, Cardone A, Orr D, Flowerday A, Katsaragakis S, Darley A, Lubowitzki S, Harris J, Skene S, Miller M, Moore M, Lewis L, DeSouza N, Donnan PT. Real time remote symptom monitoring during chemotherapy for cancer: European multicentre randomised controlled trial (eSMART). BMJ. 2021 Jul 21;374:n1647. doi: 10.1136/bmj.n1647. PMID 34289996
- [Derived] Maguire R, Fox PA, McCann L, Miaskowski C, Kotronoulas G, Miller M, Furlong E, Ream E, Armes J, Patiraki E, Gaiger A, Berg GV, Flowerday A, Donnan P, McCrone P, Apostolidis K, Harris J, Katsaragakis S, Buick AR, Kearney N. The eSMART study protocol: a randomised controlled trial to evaluate electronic symptom management using the advanced symptom management system (ASyMS) remote technology for patients with cancer. BMJ Open. 2017 Jun 6;7(5):e015016. doi: 10.1136/bmjopen-2016-015016. PMID 28592577